CLINICAL TRIAL: NCT03548584
Title: A Phase 3, 12-Week, Multicenter, Randomized, Double-blind, Placebo-controlled, 2-Arm, Fixed-dose Trial to Evaluate the Efficacy, Safety, and Tolerability of Brexpiprazole (OPC-34712) in the Treatment of Subjects With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: A Trial to Evaluate the Safety, Efficacy, and Tolerability of Brexpiprazole in Treating Agitation Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-14-213
Record Dates: First submitted 2018-05-07; First posted 2018-06-07 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Agitation Associated With Alzheimer's Dementia; Alzheimer Dementia
Keywords: Agitation
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brexpiprazole 2 mg (Experimental): Participants followed a titration schedule, to gradually increase their dose from 0.5 milligrams per day (mg/day) in the starting to 2 mg/day from Day 15. Participants continued to receive brexpiprazole 2 milligrams (mg), once daily until Week 12.
  Interventions: Drug: Brexpiprazole
- Brexpiprazole 3 mg (Experimental): Participants followed a titration schedule, to gradually increase their dose from 0.5 mg/day in the starting to 3 mg/day from Day 29. Participants continued to receive brexpiprazole 3 mg, once daily until Week 12.
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Participants received matching placebo, once daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Oral tablets
  Other Names: OPC-34712
  Arms: Brexpiprazole 2 mg; Brexpiprazole 3 mg
Other: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
This study compares the efficacy of 2 doses of brexpiprazole with placebo in participants with agitation associated with dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
This is a phase 3, 12-week, multicenter, randomized, double-blind, placebo-controlled, fixed-dose trial designed to assess the efficacy, safety, and tolerability of brexpiprazole compared with placebo. The trial consists of a 12-week double-blind treatment period with a 30 day follow-up. The trial population will include male and female participants between 55 and 90 years of age (inclusive) with a diagnosis of probable Alzheimer's disease, who are residing either in an institutionalized setting or in a non-institutionalized setting where the participant is not living alone. This trial will analyze data gathered from approximately 330 participants at multiple countries. Participants may also be eligible to enter an active treatment extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of probable Alzheimer's disease.
* Participants with a diagnosis of agitation
* Participants with a MMSE score of 5 to 22, inclusive, at screening and baseline visits.
* Participants with a previous MRI or CT scan of the brain, that was performed after the onset of symptoms of dementia, with findings consistent with a diagnosis of Alzheimer's disease.
* Participants who are residing at their current location for at least 28 days before screening and are expected to remain at the same location for the duration of the trial.
* Institutionalized participants with an identified caregiver who has sufficient contact (minimum of 2 hours per day for 4 days per week) to describe the participant's symptoms and has direct observation of the participant's behavior. Non-institutionalized participants may not be living alone and must have an identified caregiver who has sufficient contact (minimum of 2 hours per day for 4 days per week) to describe the participant's symptoms and has direct observation of the participant's behavior.
* Participants with onset of symptoms of agitation at least 2 weeks prior to screening visit.
* Participants will and able to discontinue all prohibited concomitant medications to meet protocol required washouts prior to and during the trial period.

Exclusion Criteria:

* Participants with dementia or other memory impairment not due to Alzheimer's disease.
* Participants with a history of stroke, well-documented transient ischemic attack, or pulmonary or cerebral embolism.
* Participants who had an insufficient response, based on the investigator's judgment, to 2 or more previous antipsychotic medications.
* Participants who have been diagnosed with an Axis I disorder.
* Participants who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, gastrointestinal, or psychiatric disorders.
* Participants with uncontrolled hypertension or symptomatic hypotension, or orthostatic hypotension.
* Participants with diabetes mellitus (insulin-dependent and non-insulin-dependent) may be eligible for the trial if their condition is stable and well-controlled.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Cummings JL, Chumki SR, Chang D, Zhang Z, Brubaker M, Hefting N, Such P, Wang D, Grossberg GT. Efficacy of Brexpiprazole in Participants with Agitation Associated with Dementia Due to Alzheimer's Disease: Pooled Analysis of Randomized Controlled Trials. Clin Drug Investig. 2026 Jan 27. doi: 10.1007/s40261-025-01517-9. Online ahead of print. PMID 41591746
- [Derived] Shah A, Kalu U, Chen D, Slomkowski M, Hobart M, Such P, Grossberg GT. Brexpiprazole side-effect profile in people with agitation in Alzheimer's dementia: a plain language summary. Curr Med Res Opin. 2026 Jan 14:1-3. doi: 10.1080/03007995.2025.2608578. Online ahead of print. PMID 41533472
- [Derived] Grossberg GT, Sabbagh MN, Chumki SR, Wang D, Such P, Zhang Z, Palma AM, Cummings JL. Efficacy of Brexpiprazole on Neuropsychiatric Symptoms and Impact on Caregivers: Pooled Neuropsychiatric Inventory (NPI) Analysis in Patients With Agitation Associated With Dementia due to Alzheimer's Disease. J Geriatr Psychiatry Neurol. 2025 Dec 24:8919887251407124. doi: 10.1177/08919887251407124. Online ahead of print. PMID 41439450
- [Derived] Stroud J, Cummings JL, Chumki SR, Such P, Wang D, Palma AM, Zhang Z, Brubaker M, Grossberg GT. Brexpiprazole for agitation in clinically relevant patient subgroups: a post hoc analysis of efficacy and safety in patients with agitation associated with dementia due to Alzheimer's disease. Curr Med Res Opin. 2025 Aug;41(8):1523-1534. doi: 10.1080/03007995.2025.2552278. Epub 2025 Sep 5. PMID 40847656
- [Derived] Shah A, Estilo A, Sheridan PL, Kalu U, Chen D, Chang D, Slomkowski M, Lee D, Hefting N, Hobart M, Behl S, Such P, Brubaker M, Grossberg GT. Safety and Tolerability of Brexpiprazole in Participants with Agitation Associated with Dementia due to Alzheimer's Disease: Pooled Analysis of Three Randomized Trials and an Extension Trial. CNS Drugs. 2025 Oct;39(10):1011-1023. doi: 10.1007/s40263-025-01200-9. Epub 2025 Jul 19. PMID 40681915
- [Derived] Meunier J, Creel K, Loubert A, Larsen KG, Aggarwal J, Hefting N, Oberdhan D. Defining a clinically meaningful within-patient change threshold for the Cohen-Mansfield Agitation Inventory in Alzheimer's dementia. Front Neurol. 2024 Jul 23;15:1379062. doi: 10.3389/fneur.2024.1379062. eCollection 2024. PMID 39108660
- [Derived] Lee D, Slomkowski M, Hefting N, Chen D, Larsen KG, Kohegyi E, Hobart M, Cummings JL, Grossberg GT. Brexpiprazole for the Treatment of Agitation in Alzheimer Dementia: A Randomized Clinical Trial. JAMA Neurol. 2023 Dec 1;80(12):1307-1316. doi: 10.1001/jamaneurol.2023.3810. PMID 37930669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 345 participants were randomized, and participated in the study from 16 May 2018 to 1 June 2022.
Period: Overall Study
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 3 mg | Placebo
Started | 75 | 153 | 117
Intent-to-treat Population (Intent-to-treat (ITT) Population consisted of all participants in the randomized sample, who took at least 1 dose of investigational medical product (IMP) and had a baseline and at least one post-baseline evaluation for the Cohen-Mansfield Agitation Inventory (CMAI) total score.) | 73 | 153 | 116
Completed | 68 | 130 | 104
Not Completed | 7 | 23 | 13
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 1 | 11 | 5
Not completed — Site Terminated by Sponsor | 1 | 3 | 2
Not completed — Subject Withdrew Consent to Participate | 5 | 5 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Non-compliance with Study Drug | 0 | 1 | 0
Not completed — Reason not Specified (Not Related to Coronavirus Disease 2019 [COVID-19]) | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Sample consisted of all participants who were randomized into this trial.
Groups:
- Brexpiprazole 2 mg: Participants followed a titration schedule, to gradually increase their dose from 0.5 mg/day in the starting to 2 mg/day from Day 15. Participants continued to receive brexpiprazole 2 mg, once daily until Week 12.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 3 mg | Placebo | Total
Number analyzed (Participants) | 75 | 153 | 117 | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (7.3) | 74.6 (8.0) | 73.0 (7.0) | 74.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 92 | 60 | 195
  Male | 32 | 61 | 57 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 46 | 37 | 108
  Not Hispanic or Latino | 50 | 107 | 80 | 237
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 1 | 12
  White | 70 | 144 | 115 | 329
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Cohen-Mansfield Agitation Inventory (CMAI) Total Score [Mean (Standard Deviation); unit: score on a scale] — The CMAI assesses frequency of agitated behaviors in elderly persons. The scale consists of 29 agitated behaviors that are further categorized into distinct agitation syndromes, also known as CMAI factors of agitation. Each of the agitated behaviors are scored 1 (never) to 7 (several times an hours), with the total scale score ranging from 29 to 203. Higher score indicates greater frequency of agitated behavior.
  score on a scale | 78.6 (15.5) | 81.2 (17.2) | 79.4 (17.6) | 80 (17)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the CMAI Total Score
Description: The CMAI score is used to assess the frequency of manifestations of agitated behaviors in participants. The CMAI consists of 29 agitated behaviors that are rated on a 7-point scale of frequency across four subscales of aggressive behavior, physically nonaggressive behavior, verbally agitated behavior and hiding and hoarding as: 1=never; 2=less than once a week; 3=once or twice a week; 4=several times a week; 5=once or twice a day; 6=several times a day; 7=several times an hour. The CMAI total score ranges from 29 to 203. Higher scores indicate worsening of the condition. A negative change from baseline indicates improvement. Mixed model repeated measures (MMRM) was used for the analysis. As prespecified in the statistical analysis plan (SAP), data for this outcome measure was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Time Frame: Baseline and Week 12
Population: The ITT Population consisted of all participants in the randomized sample, who took at least 1 dose of IMP and had a baseline and at least one post-baseline evaluation for the CMAI total score. Overall number analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Brexpiprazole 2 and 3 mg: Participants followed a titration schedule, to gradually increase their dose from 0.5 mg/day in the starting to 2 mg/day from Day 15 or from 0.5 mg/day in the starting to 3 mg/day from Day 29.
  Participants continued to receive brexpiprazole 2 or 3 mg, once daily until Week 12.
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
score on a scale | -22.6 (1.08) | -17.3 (1.44)
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Test type: Superiority; p = 0.0026, MMRM — MMRM method with model terms of treatment, trial site, visit, treatment-by-visit and baseline-by-visit interaction were used for analysis; LS Mean Difference = -5.32, 95% CI 2-sided [-8.77 to -1.87]

2. Secondary Outcome: Change From Baseline to Week 12 in the Clinical Global Impression Severity of Illness (CGI-S) Score, as Related to Agitation
Description: CGI-S was used to rate the severity of agitation. The score ranges from 0 to 7 with response choices as, 0=not assessed; 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. The higher the value, the more severe the agitation. A negative change from baseline indicates improvement. MMRM was used for the analysis. As prespecified in the SAP, data for this outcome measure was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
score on a scale | -1.20 (0.06) | -0.93 (0.08)
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Test type: Superiority; p = 0.0078, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.47 to -0.07]

3. Secondary Outcome: Change From Baseline to Week 12 in CMAI Subscale Scores
Description: The CMAI score is used to assess the frequency of manifestations of agitated behaviors in participants. It consists of 29 agitated behaviors that are rated on a 7-point scale of frequency across four subscales of aggressive behavior, physically nonaggressive behavior, verbally agitated behavior and hiding and hoarding, as: 1=never; 2=less than once a week; 3=once or twice a week; 4=several times a week; 5=once or twice a day; 6=several times a day; 7=several times an hour. The four subscales include 12, 6, 4, and 2 items, respectively. The score of the subscale is the sum of the individual items included in the subscale, so the score range for each of the 4 subscales is 0 to 84, 0 to 42, 0 to 28, and 0 to 14, respectively. Higher scores indicate worsening of the condition. A negative change from baseline=improvement. MMRM was used for the analysis. As prespecified in the SAP, data for this outcome measure was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
score on a scale
  Aggressive Behavior | -9.09 (0.42) | -7.13 (0.56)
  Physically Nonaggressive Behavior | -6.45 (0.40) | -5.04 (0.53)
  Verbally Agitated Behavior | -4.39 (0.31) | -3.14 (0.40)
  Hiding and Hoarding | -1.50 (0.17) | -1.14 (0.23)
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Aggressive Behavior; Test type: Superiority; p = 0.0040, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.95, 95% CI 2-sided [-3.28 to -0.63]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Physically Nonaggressive Behavior; Test type: Superiority; p = 0.0296, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.41, 95% CI 2-sided [-2.68 to -0.14]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Verbally Agitated Behavior; Test type: Superiority; p = 0.0113, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.24, 95% CI 2-sided [-2.21 to -0.28]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Hiding and Hoarding; Test type: Superiority; p = 0.1941, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.36, 95% CI 2-sided [-0.90 to 0.18]

4. Secondary Outcome: Change From Baseline in CMAI Total Score for Each Trial Visit During the Double-blind Treatment Period
Description: The CMAI score is used to assess the frequency of manifestations of agitated behaviors in participants. The CMAI consists of 29 agitated behaviors that are rated on a 7-point scale of frequency across four subscales of aggressive behavior, physically nonaggressive behavior, verbally agitated behavior and hiding and hoarding as: 1=never; 2=less than once a week; 3=once or twice a week; 4=several times a week; 5=once or twice a day; 6=several times a day; 7=several times an hour. The CMAI total score ranges from 29 to 203. Higher scores indicate worsening of the condition. A negative change from baseline indicates improvement. MMRM was used for the analysis. As prespecified in the SAP, data for this outcome measure was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
score on a scale
  Change From Baseline at Week 2 | -5.76 (0.71) | -6.61 (0.90)
  Change From Baseline at Week 4 | -12.1 (0.82) | -11.0 (1.06)
  Change From Baseline at Week 6 | -16.2 (0.91) | -13.9 (1.19)
  Change From Baseline at Week 8 | -19.4 (0.96) | -14.4 (1.28)
  Change From Baseline at Week 10 | -22.2 (0.97) | -15.7 (1.29)
  Change From Baseline at Week 12 | -22.6 (1.08) | -17.3 (1.44)
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change From Baseline at Week 2; Test type: Superiority; p = 0.4242, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.85, 95% CI 2-sided [-1.24 to 2.93]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change From Baseline at Week 4; Test type: Superiority; p = 0.3665, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.14, 95% CI 2-sided [-3.63 to 1.34]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 6; Test type: Superiority; p = 0.1065, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -2.32, 95% CI 2-sided [-5.15 to 0.50]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 8; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -5.08, 95% CI 2-sided [-8.12 to -2.05]
Statistical Analysis 5: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 10; Test type: Superiority; p < .0001, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -6.47, 95% CI 2-sided [-9.54 to -3.40]
Statistical Analysis 6: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 12; Test type: Superiority; p = 0.0026, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -5.32, 95% CI 2-sided [-8.77 to -1.87]

5. Secondary Outcome: Change From Baseline in CGI-S for Each Trial Visit During the Double-Blind Treatment Period
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
score on a scale
  Change From Baseline at Week 2 | -0.21 (0.03) | -0.27 (0.04)
  Change From Baseline at Week 4 | -0.53 (0.05) | -0.50 (0.06)
  Change From Baseline at Week 6 | -0.74 (0.05) | -0.68 (0.07)
  Change From Baseline at Week 8 | -0.97 (0.06) | -0.70 (0.08)
  Change From Baseline at Week 10 | -1.14 (0.06) | -0.86 (0.08)
  Change From Baseline at Week 12 | -1.20 (0.06) | -0.93 (0.08)
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 2; Test type: Superiority; p = 0.3048, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.05, 95% CI 2-sided [-0.05 to 0.16]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 4; Test type: Superiority; p = 0.7058, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.03, 95% CI 2-sided [-0.17 to 0.12]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 6; Test type: Superiority; p = 0.4516, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.06, 95% CI 2-sided [-0.23 to 0.10]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 8; Test type: Superiority; p = 0.0052, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.46 to -0.08]
Statistical Analysis 5: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 10; Test type: Superiority; p = 0.0060, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.47 to -0.08]
Statistical Analysis 6: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Change from Baseline at Week 12; Test type: Superiority; p = 0.0078, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.47 to -0.07]

6. Secondary Outcome: Clinical Global Impressions-Improvement (CGI-I) Score at Each Trial Visit During the Double-Blind Treatment Period
Description: CGI-I is a 7-point scale that requires the clinician to assess whether a participant's condition has improved or worsened relative to a baseline state at the beginning of the intervention. This was rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; or 7=very much worse. Higher scores indicate worse condition. As prespecified in the SAP, data for this outcome measure was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 12
Population: The ITT Population consisted of all participants in the randomized sample, who took at least 1 dose of IMP and had a baseline and at least one post-baseline evaluation for the CMAI total score. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
score on a scale
  Week 2: number analyzed (Participants) | 221 | 114
  Week 2 | 3.70 (0.75) | 3.57 (0.69)
  Week 4 | 3.19 (0.85) | 3.39 (0.87)
  Week 6 | 2.92 (0.94) | 3.19 (0.95)
  Week 8 | 2.80 (1.00) | 3.16 (1.01)
  Week 10 | 2.62 (0.99) | 2.97 (1.00)
  Week 12 | 2.66 (1.09) | 2.97 (1.12)
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1975, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.05 to 0.26]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0084, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.44 to -0.06]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0101, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.46 to -0.06]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 8; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.59 to -0.15]
Statistical Analysis 5: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0023, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.55 to -0.12]
Statistical Analysis 6: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0070, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.57 to -0.09]

7. Secondary Outcome: CMAI Response Rate Assessed as Percentage of Participants With CMAI Response at Every Scheduled Trial Visit in the Double-Blind Treatment Period
Description: The CMAI assesses frequency of agitated behaviors in elderly persons. The scale consists of 29 agitated behaviors that are further categorized into distinct agitation syndromes, also known as CMAI factors of agitation. Each of the agitated behaviors are scored 1 (never) to 7 (several times an hours), with the total scale score ranging from 29 to 203. Higher score indicates greater frequency of agitated behavior. As prespecified in the SAP, data for this outcome measure was analyzed and reported in a combined way for brexpiprazole 2 and 3 mg.
Time Frame: Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
percentage of participants
  >/= 20%: Week 2: number analyzed (Participants) | 221 | 114
  >/= 20%: Week 2 | 11.3 | 13.2
  >/= 20%: Week 4 | 29.3 | 27.6
  >/= 20%: Week 6 | 43.1 | 37.9
  >/= 20%: Week 8 | 59.6 | 38.8
  >/= 20%: Week 10 | 65.8 | 45.7
  >/= 20%: Week 12 | 68.4 | 47.4
  >/= 30%: Week 2: number analyzed (Participants) | 221 | 114
  >/= 30%: Week 2 | 3.62 | 3.51
  >/= 30%: Week 4 | 10.7 | 10.3
  >/= 30%: Week 6 | 22.7 | 20.7
  >/= 30%: Week 8 | 32.9 | 19.0
  >/= 30%: Week 10 | 38.2 | 24.1
  >/= 30%: Week 12 | 42.7 | 25.9
  >/= 40%: Week 2: number analyzed (Participants) | 221 | 114
  >/= 40%: Week 2 | 1.81 | 1.75
  >/= 40%: Week 4 | 4.89 | 5.17
  >/= 40%: Week 6 | 10.7 | 8.62
  >/= 40%: Week 8 | 16.9 | 8.62
  >/= 40%: Week 10 | 20.9 | 11.2
  >/= 40%: Week 12 | 23.1 | 14.7
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/= 20%: Week 2; Test type: Superiority; p = 0.7290, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.10, 95% CI 2-sided [0.64 to 1.91]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=20%: Week 4; Test type: Superiority; p = 0.6196, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.09, 95% CI 2-sided [0.78 to 1.52]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=20%: Week 6; Test type: Superiority; p = 0.2718, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.16, 95% CI 2-sided [0.88 to 1.53]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=20%: Week 8; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.52, 95% CI 2-sided [1.19 to 1.93]
Statistical Analysis 5: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=20%: Week 10; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.42, 95% CI 2-sided [1.15 to 1.76]
Statistical Analysis 6: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=20%: Week 12; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.41, 95% CI 2-sided [1.15 to 1.72]
Statistical Analysis 7: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=30%: Week 2; Test type: Superiority; p = 0.7211, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.22, 95% CI 2-sided [0.39 to 3.85]
Statistical Analysis 8: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=30%: Week 4; Test type: Superiority; p = 0.7606, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.11, 95% CI 2-sided [0.57 to 2.14]
Statistical Analysis 9: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=30%: Week 6; Test type: Superiority; p = 0.5902, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.12, 95% CI 2-sided [0.74 to 1.68]
Statistical Analysis 10: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=30%: Week 8; Test type: Superiority; p = 0.0054, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.70, 95% CI 2-sided [1.14 to 2.54]
Statistical Analysis 11: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=30%: Week 10; Test type: Superiority; p = 0.0066, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.59, 95% CI 2-sided [1.11 to 2.26]
Statistical Analysis 12: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=30%: Week 12; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.62, 95% CI 2-sided [1.18 to 2.23]
Statistical Analysis 13: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=40%: Week 2; Test type: Superiority; p = 0.9074, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.11, 95% CI 2-sided [0.20 to 5.97]
Statistical Analysis 14: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=40%: Week 4; Test type: Superiority; p = 0.9625, Cochran-Mantel-Haenszel; Ratio of Response Rate = 0.98, 95% CI 2-sided [0.36 to 2.64]
Statistical Analysis 15: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=40%: Week 6; Test type: Superiority; p = 0.5120, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.26, 95% CI 2-sided [0.63 to 2.53]
Statistical Analysis 16: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=40%: Week 8; Test type: Superiority; p = 0.0244, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.98, 95% CI 2-sided [1.03 to 3.79]
Statistical Analysis 17: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=40%: Week 10; Test type: Superiority; p = 0.0161, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.86, 95% CI 2-sided [1.08 to 3.18]
Statistical Analysis 18: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; >/=40%: Week 12; Test type: Superiority; p = 0.0347, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.62, 95% CI 2-sided [1.00 to 2.61]

8. Secondary Outcome: CMAI Response Rate Assessed as Percentage of Participants With CMAI Response Based on Improvement From Baseline in Agitation Status at Every Scheduled Trial Visit in the Double-Blind Treatment Period
Description: as for outcome 7
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
percentage of participants
  Week 2: number analyzed (Participants) | 221 | 114
  Week 2 | 8.14 | 14.0
  Week 4 | 20.4 | 19.0
  Week 6 | 33.8 | 26.7
  Week 8 | 44.0 | 31.0
  Week 10 | 50.2 | 34.5
  Week 12 | 52.4 | 37.1
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1503, Cochran-Mantel-Haenszel; Ratio of Response Rate = 0.64, 95% CI 2-sided [0.35 to 1.16]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 4; Test type: Superiority; p = 0.7559, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.07, 95% CI 2-sided [0.69 to 1.67]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 6; Test type: Superiority; p = 0.2246, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.23, 95% CI 2-sided [0.88 to 1.72]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 8; Test type: Superiority; p = 0.0276, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.38, 95% CI 2-sided [1.02 to 1.87]
Statistical Analysis 5: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0031, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.46, 95% CI 2-sided [1.12 to 1.89]
Statistical Analysis 6: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.47, 95% CI 2-sided [1.14 to 1.89]

9. Secondary Outcome: CGI-I Response Rate Assessed as Percentage of Participants With CGI-I Response at Every Scheduled Trial Visit in the Double-Blind Treatment Period
Description: as for outcome 6
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole 2 and 3 mg | Placebo
Number analyzed (Participants) | 225 | 116
percentage of participants
  Week 2: number analyzed (Participants) | 221 | 114
  Week 2 | 4.98 | 5.26
  Week 4 | 21.8 | 12.1
  Week 6 | 35.1 | 23.3
  Week 8 | 44.4 | 24.1
  Week 10 | 52.4 | 33.6
  Week 12 | 52.4 | 40.5
Statistical Analysis 1: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 2; Test type: Superiority; p = 0.8549, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.10, 95% CI 2-sided [0.40 to 3.03]
Statistical Analysis 2: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 4; Test type: Superiority; p = 0.0093, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.95, 95% CI 2-sided [1.14 to 3.32]
Statistical Analysis 3: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0083, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.56, 95% CI 2-sided [1.10 to 2.22]
Statistical Analysis 4: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 8; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.85, 95% CI 2-sided [1.32 to 2.58]
Statistical Analysis 5: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.57, 95% CI 2-sided [1.18 to 2.09]
Statistical Analysis 6: Comparison: Brexpiprazole 2 and 3 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0160, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.32, 95% CI 2-sided [1.03 to 1.69]

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to end of study (Week 16)
Description: Randomized Sample was used to assess all-cause mortality. It consisted of all participants who were randomized into this trial. Safety Sample was used to assess serious adverse events (SAEs) and other adverse events (AEs) and consisted of all participants who were administered at least one dose of IMP.
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 3 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 1/153 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/73 | 6/153 | 3/116
Other Adverse Events (participants affected / at risk) | 5/73 | 10/153 | 8/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2 mg (N=73) | Brexpiprazole 3 mg (N=153) | Placebo (N=116)
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sars-Cov-2 test positive (Investigations) | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Mental status change (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2 mg (N=73) | Brexpiprazole 3 mg (N=153) | Placebo (N=116)
Headache (Nervous system disorders) | 5 | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT03548584/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03548584/SAP_001.pdf